CLINICAL TRIAL: NCT03616275
Title: Improving the Glycemic Regulation and the Psychoneuroimmunological Function by Enhancing the Vagal Tone in Prediabetes Individuals
Brief Title: Enhancing the Vagal Tone in Prediabetes Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Yu-Ju Chen, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2-106-05005
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Prediabetes; Autonomic Nervous System Imbalance; Poor Glycemic Control; Psychological Distress
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRV biofeedback group (Experimental): 8 once-a-week, individual, 30-min sessions of HRV biofeedback and 1 session of healthy lifestyle education
  Interventions: Other: HRV biofeedback
- control group (No Intervention): 1 session of healthy lifestyle education

INTERVENTIONS:
Other: HRV biofeedback — HRV biofeedback protocol is modified from Lehrer's HRV biofeedback manual (2000), which had been successfully used to improve functioning and quality of life for patients with asthma and COPD. A noninvasive biofeedback system with a NeXus-10 with BioTrace+ (Mind Media B.V., Netherlands) and laptop computer will be used for biofeedback intervention. The intervention protocol is including paced breathing in resonant frequency, abdominal breathing and pursed-lip breathing, and visual biofeedback. The designed intervention protocol will include 8 once-a-week, individual, 20-min in hospital training sessions and twice-a-day, 20-min home self-practices.
  Arms: HRV biofeedback group

SUMMARY:
This is a 2-year course of study. A randomized control trial will be conducted, in which 90 prediabetes individuals will be recruited and randomly assigned them into the wait-list control group or experimental group to test the effectiveness of 8 once-a-week, individual, 20-min sessions of HRV biofeedback on modulating vagal tone, glycemic control, psychological wellbeing, and inflammatory status in this population. Its longitudinal effects will be evaluated after 3- and 6-month follow-up.

DETAILED DESCRIPTION:
Background. Compared to healthy population, individuals with prediabetes have a higher risk to develop diabetes and other cardiovascular diseases. However, these downward progressions might positively associate with autonomic nervous dysfunction, especially low vagal tone, which can be detected prior to comorbidities confirmed. The significant correlations among low autonomic nervous, high psychological distress, inflammatory status, and poor glycemic regulation, which are regarded as the psychoneuroimmunological integration, have not been well studied in prediabetes individuals. Heart rate variability (HRV) biofeedback is an easy and noninvasive intervention, which has been confirmed to strengthen baroreflex stimulation, facilitate the modulation of vagal tone, and further promote the physiological and psychological wellbeing in various diseases but not in prediabetes.

Objective. To test the effectiveness of HRV biofeedback on the modulating vagal tone and further enhancing the psychoneuroimmunological integration related to glycemic control, anti-inflammatory reaction, and psychological wellbeing.

Research methods. In this 2-year RCT study, the investigators are planning to recruit 90 prediabetes individuals and randomly assigned them into wait-list control group or experimental group by using the random sequence of numbers generated from the Excel Bernoulli Function. Experimental group will receive 8 once-a-week, individual, 30-min sessions of HRV biofeedback and 1 session of healthy lifestyle education. During the biofeedback training period, subjects will be encouraged to self- home practice of resonant frequency breathing for 20 mins, twice-a-day. Control group will receive 1 session of healthy lifestyle education. All subjects will be repeatedly assessed at time of enrollment, post-training (8 weeks after enrollment), 3-month, and 6-month follow-up. Repeated assessments will include physiological measurements of HRV, BDNF, GAS6, HbA1c, CRP, IL- 6, FPG, and salivary cortisol, and psychological measurements of perceived stress, anxiety, and depression.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 or more
* fasting blood glucose level of 100 to 125 mg/dl
* HbA1C value of 5.7% to 6.4%

Exclusion Criteria:

* lack of Chinese literacy
* visual and hearing deficits
* the presence of arrhythmia
* previous diagnosed with diabetes
* any other serious physical illness (e.g. severe neurocognitive disorders or evidence of cor pulmonale) or psychiatric disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline Autonomic function (Heart rate variability) at 3 and 6 months | baseline, 3-month, and 6-month visits
  Heart rate variability (HRV) was used to represent the autonomic function, and measured with Mind Media B.V. (NeXus-10, Netherlands). Time and frequency domains of HRV was analyzed using Kubios HRV software (Biosignal Analysis and Medical Imaging Group, Finland).

SECONDARY OUTCOMES:
Changes from Baseline Psychological distress (Anxiety and Depression) at 3 and 6 months | baseline, 3-month, and 6-month visits
  The hospital anxiety and depression scale was a 14-item ordinal scale, used for participants to self-rate their psychological distress related to anxiety (7 items) and depression (7 items). Items are scored 0(no distress) to 3 (serious distress). Based on the findings from previous studies, scoring at or higher than the cut-off point of 8 out of 21, identified those with anxiety or depression.
Changes from Baseline perceived stress at 3 and 6 months | baseline, 3-month, and 6-month visits
  Perceived stress was measured using the Chinese version of the Perceived Stress Scale (PSS), through which the participants self-reported about how they cope with, react to, and feel about various stressors. The PSS is a 5-point scale that ranges from 0 (never) to 4 (very often) with 14 items (seven negative and seven positive).
Changes from Baseline serum biomarkers (CRP, IL-6, BDNF, GAS6, HbA1c, and FPG) at 3 and 6 months | baseline, 3-month, and 6-month visits
  All blood will be drawn in the morning, between 8 and 10 a.m., and will immediately be separated by centrifugation at 2000 r/min for 10 minutes at 4 oC. CRP, BDNF, and GAS6 will be measured with a sandwich enzyme-linked immunoassay (ELISA) using a DuoSet ELISA Development kit (R&D Systems Catalog # DY1707). IL-6 will be measured by the BD™ CBA Human Soluble Protein Flex Set System with discrete fluorescence intensities to detect soluble analytes at very low concentrations. The HbA1c value will be measured by high-performance liquid chromatography, using the Primus CLC385 (Primus Corporation, Kansas City, MO). The FPG will be measured using a Reflotron reflectance photometric analyzer (Boehringer Mannheim, Germany).
Changes from Baseline salivary cortisol at 3 and 6 months | baseline, 3-month, and 6-month visits
  Participant will be requested to collect the saliva before breakfast, approximately 30 minutes after awakening and before they brushed their teeth. The sample will be immediately frozen and transported to the laboratory for cortisol concentration measurement and analyzed using a commercial ELISA kit (Calbiochem, Darmstadt, Germany). All salivary variables are normalized by salivary flow rate.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ju Chen, Ph.D., Principal Investigator — National Defense Medical Center, Taiwan
Locations (1):
- Tri-Service Medical Center, Taipei, Taiwan